CLINICAL TRIAL: NCT00550758
Title: The Effect of Singular (Montelukast) 4mg on Hypersensitivity of the Airways in Children 3-5 Years Old. + Extended Study Hyprsensitivity of the Airways in Asthmatic Children Age 3-6years
Brief Title: Spirometry and Methacholine Challenge Test in Asthmatic Children Age 3-6years
Acronym: MCH-preschool
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the study has recently ended, all information gathred as planed
Sponsor: Rambam Health Care Campus (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: McH-Spir- preschool_CTIL
Record Dates: First submitted 2007-10-20; First posted 2007-10-30 (Estimated); Last update posted 2007-10-30 (Estimated); Status verified 2007-10

CONDITIONS: Asthma; Recurrent Cough
Keywords: Methacholine challenge; Spirometry, Early childhood
MeSH Terms: conditions — Asthma; Cough | interventions — Spirometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Methachoine — inhalation of triple-concentration increments (0.06 to13.9mg/ml/methacholine)
Device: spirometry — spirometry

SUMMARY:
Rational: The possible contribution of methacholine challenge test via spirometry to the clinical diagnosis of young children with various respiratory symptoms, the most appropriate spirometry index, and the proper cutoff point concentration that will define airway sensitivity have not yet been explored. Objectives: To assess airway reactivity by spirometry in a large group of children aged 3-6years with various respiratory symptoms.

DETAILED DESCRIPTION:
We aimed to gather information concerning methacholine challenge test performed in children previously diagnosed with asthma (asthmatics) and 48 had prolonged cough (coughers) from the pediatric clinic at Meyer Children's Hospital.

Tests were performed by inhalation of triple-concentration increments (0.06 to13.9mg/ml/methacholine).

Spirometry was determined at baseline and after each inhalation in duplicate sets. End of test was defined by a fall of 20%FEV1 baseline (PC20-FEV1). PC20-FEV1<4.0mg/ml was considered positive). Results from the challenge were related to data from questionnaires concerning respiratory symptoms were analyzed at the end of the studies.

ELIGIBILITY:
Inclusion Criteria:

* age 3- to 6-years
* respiratory diseases who were highly indicative of asthma diagnosis according to GINA guidelines [9]
* cough duration of more than 4 weeks
* normal chest auscultation and baseline FEV1>75% predicted for healthy preschool children, on the day of testing.

Exclusion Criteria:

* presence of other chronic respiratory conditions
* emergency room visit or the presence of respiratory infection within the last month
* oral or inhaled steroids or other anti-inflammatory medication taken in the last two weeks
* bronchodilator taken within 24-hours prior to the test.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2004-05; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Determination of a Fall of 20% FEV1 from baseline values (PC20FEV1) | after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lea Bentur, MD, Study Director — Rambam Health Care Campus; Daphna Vilozni, PhD, Principal Investigator — Rambam Health Care Campus